CLINICAL TRIAL: NCT02658539
Title: Impact of Physiological, Lifestyle and Genetic Factors on Body Composition
Acronym: BODYCON
Status: Completed | Type: Observational
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Julie Lovegrove, Prof BSc Diet (Dip) PhD RNutr FAfN, University of Reading
Other Study IDs: 13/55; 14/SC/1095 (Other: NHS Research Ethics Committee)
Record Dates: First submitted 2016-01-08; First posted 2016-01-20 (Estimated); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Body Composition, Beneficial
Keywords: Body fat distribution; Bone mineral density; Dual-energy x-ray absorptiometry
MeSH Terms: conditions — Glucocorticoid Receptor Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — A fasting blood sample will be taken at the end of the study visit for the measurement of fasting lipids (total and high density lipoprotein-cholesterol, triacylglycerol and non-esterified fatty acids), glucose, insulin, C-reactive protein and for vitamin D status.
  The buffy coat (consisting of white blood cells) will be isolated from the blood sample for genotyping analysis.
Oversight: Data Monitoring Committee: No

SUMMARY:
Research has shown that body composition is a key component of health and future disease risk. Being overweight and obese is associated with a higher body fat composition, and a greater risk of developing type II diabetes and heart disease. The location where fat is stored in the body is becoming increasingly recognised an important predictor of risk, with extra fat around the abdomen and waist (referred to as the android pattern of fat distribution or 'apple' shape) thought to increase your disease risk than storing fat around the thighs and buttocks (gynoid pattern of fat distribution or 'pear' shape). As a result, there is significant interest in techniques to accurately monitor and detect changes in body composition, and also physiological and lifestyle factors which influence body fat, lean tissue mass and bone mineral density. This cross sectional human study will look at how physiological, behavioural and genetic factors relate to total body composition in 1,196 healthy men and women aged between 18 and 70 years. Interested applicants will be invited to attend for a single visit at the Hugh Sinclair Unit of Human Nutrition at the University of Reading. This visit lasts around two hours and includes noninvasive measures of body composition (bio-electrical impedance and dual energy x-ray absorptiometry), arterial stiffness and fasting measures of metabolic health. Diet and physical activity will then be monitored over a four day period using diet and activity diaries, and an activity monitor. The findings from this study will contribute to the evidence base on how subject characteristics influence body composition and inform on the design of future human studies on body composition methodology.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5-39.9 kg/m2
* Not having suffered a myocardial infarction/stroke in the past 12 months
* Not hyperlipidaemic (total cholesterol level < 7.8 mmol/l and triacylglycerol < 2.3 mmol/l).
* Not diabetic (diagnosed as fasting blood glucose > 7 mmol/l) or suffer from other endocrine disorders
* Not suffering from renal or bowel disease or have a history of cholestatic liver disease or pancreatitis
* Not diagnosed with cancer
* Not suffering from arthritis or fracture deformity of the spine or femur
* Not undergone bone related surgeries such as hip replacement or fusion(s)
* Not on drug treatment for hyperlipidaemia, hypertension, inflammation or hypercoagulation
* No history of alcohol abuse
* Not anaemic (Haemoglobin >115 g/l for women and 125 g/l for men)

Exclusion Criteria:

Due to the use of ionising radiation by the dual energy x-ray absorptiometry (DXA) scanner to assess total body composition and bone mineral density, the following exclusion criteria apply:

* Females who are breastfeeding, may be pregnant, or if of childbearing potential and are not using effective contraceptive precautions.
* Individuals with other radio-opaque implants (such as a knee or other joint replacement) or medical devices (such as a pacemaker).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women living in and around Reading, Berkshire, United Kingdom
Sampling Method: Probability Sample
Enrollment: 370 (Actual)
Dates: Start 2016-02; Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Total body composition | 1 year
  Measured using dual-energy x-ray absorptiometry

SECONDARY OUTCOMES:
Body composition | 1 year
  Assessed using bio-electrical impedance
Fasting blood lipids | 1 year
  Total cholesterol, triacylglycerol, high density lipoprotein cholesterol, low density lipoprotein cholesterol and non-esterified fatty acids
Markers of insulin resistance | 1 year
  Glucose, insulin and indices of insulin resistance/sensitivity
Arterial stiffness | 1 year
  Stiffness index and Reflection index measured using digital volume pulse and Mobil-O-Graph
Blood pressure | 1 year
  Systolic and diastolic blood pressure
C-reactive protein | 1 year
  Measured using a clinical chemistry analyser
Dietary intake | 1 year
  Assessed using a 4-day weighed intake
Physical activity | 1 year
  Assessed over 4 days using an accelerometer and activity diary
Anthropometric measurements | 1 year
  Body mass index, waist circumference and hip circumference

OTHER OUTCOMES:
Genotyping | 1 year
  Single nucleotide polymorphisms in genes associated with body composition
Vitamin D status (25 hydroxy vitamin D) | 1 year
  Assessed using HPLC or GC-MS

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Lovegrove, BSc PhD, Principal Investigator — University of Reading
Locations (1):
- Department of Food and Nutritional Sciences, University of Reading, Reading, Berkshire, United Kingdom

REFERENCES:
- [Derived] Ozen E, Mihaylova R, Weech M, Kinsella S, Lovegrove JA, Jackson KG. Association between dietary saturated fat with cardiovascular disease risk markers and body composition in healthy adults: findings from the cross-sectional BODYCON study. Nutr Metab (Lond). 2022 Mar 3;19(1):15. doi: 10.1186/s12986-022-00650-y. PMID 35241101